CLINICAL TRIAL: NCT06208241
Title: Use of Allocetra-OTS in End Stage Knee Osteoarthritis - Assessment of Safety
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Amir Oron (Other)
Collaborators: Enlivex Therapeutics Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Amir Oron, Principal investigator, Kaplan Medical Center
Organization: Kaplan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 189-22
Record Dates: First submitted 2023-09-06; First posted 2024-01-17 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Allocetra-OTS (Experimental): Two IA dose of Allocetra-OTS cells in suspension
  Interventions: Drug: Allocetra-OTS

INTERVENTIONS:
Drug: Allocetra-OTS — Allocetra-OTS is a cell-based therapy consisting of non-HLA-matched allogeneic peripheral blood mononuclear cells, derived from a healthy human donor following a leukapheresis procedure, induced to an apoptotic stable state and suspended in a solution containing DMSO.

SUMMARY:
This is a pilot study to assess safety and possible efficacy of Allocetra-OTS in end-stage knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older.
2. Diagnosed with end-stage knee osteoarthritis and are scheduled or offered surgery.
3. X-ray positive for knee osteoarthritis.
4. Pain and functional disability from osteoarthritis.
5. Acceptable blood workup results (CBC, electrolytes, kidney and liver function) from up to three months before treatment.
6. Mentally and physically able to fully comply with the study protocol.
7. Signed Informed Consent form.

Exclusion Criteria:

1. Evidence of active local infection in the vicinity of the knee joint.
2. Previous surgery of total or partial knee replacement in the injected knee.
3. Patients unable to provide informed consent due to language barrier or mental status.
4. Patients with a major medical condition that would affect quality of life and influence the results of the study.
5. Patients unwilling to be followed for the duration of the study.
6. Acute infection requiring intravenous antibiotics at the time of screening.
7. Other limb pain of unknown etiology.
8. Pain in the limb clinically assessed to arise from an origin which is not the affected knee joint.
9. Known neurological disease or rheumatic condition other than osteoarthritis.
10. Bleeding disorders.
11. Known cognitive disorder.
12. Concurrent participation in any other clinical study. Participation in an interventional investigational study within 30 days prior to enrollment.
13. Physician objection.
14. Positive pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events and Serious adverse events following Allocetra-OTS injection | 6 months
  The safety and tolerability endpoint evaluates the incidence and severity of complications following intraarticular injection of Allocetra-OTS:
  * Injection-related reactions occurring during Allocetra-OTS injection, including injection interruption/discontinuation.
  * Treatment-emergent adverse events following Allocetra-OTS injection.
  * Treatment-emergent serious adverse events.
  * Adverse events or serious adverse events related to the use of Allocetra-OTS as an intraarticular injection material.
  * Safety assessments beyond 1 month following injection will focus on events that are at least possibly related to Allocetra-OTS treatment.

SECONDARY OUTCOMES:
Efficacy of Allocetra-OTS- Pain mitigation as measured by Visual Analog Scale tool. | 6 months
  To assess the efficacy of Allocetra-OTS. Secondary endpoints for efficacy will be measured in terms of:
  • Pain mitigation as measured by VAS (Visual Analog Scale) tool in a range of 0-10 points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) response change along study period | 6 month
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) response change along study period (questionnaires aimed at assessing arthritis related function ).
  The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
SF-36 questionnaire response change along study period | 6 month
  SF-36 questionnaire response change along study period (questionnaires aimed at assessing quality of life,).

CONTACTS AND LOCATIONS:
Overall Officials: Amir Oron, MD, Principal Investigator — Kaplan Medical Center
Locations (1):
- Kaplan Medical Center, Rehovot, Israel